CLINICAL TRIAL: NCT04072146
Title: Open-Label, Single-Center, Randomized, 2-way Crossover Study Evaluating Relative Bioavailability of OC-01 (Varenicline) Nasal Spray as Compared to Orally Administered Varenicline (the Zen Study)
Brief Title: Evaluating Relative Bioavailability of OC-01 (Varenicline) Nasal Spray as Compared to Orally Administered Varenicline
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Oyster Point Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: OPP-100
Record Dates: First submitted 2019-08-27; First posted 2019-08-28 (Actual); Results first posted 2022-05-23 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — Nasal Sprays; Varenicline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Varenicline oral tablet 1mg, then OC-01 (varenicline solution) nasal spray 0.12 mg (Experimental): OC-01 0.12 mg was administered intranasally 50 ul into each nostril in a fasted state
  Interventions: Drug: Vaenicline oral tablet 1 mg, then OC-01 (varenicline solution) nasal spray 0.12 mg
- OC-01 (varenicline solution) nasal spray 0.12 mg, then Varenicline oral tablet 1 mg (Active Comparator): Varenicline oral tablet 1mg was administered orally in a fasted stated with 200 ml water
  Interventions: Drug: OC-01 (varenicline solution) nasal spray 0.12 mg then Varenicline oral tablet 1 mg

INTERVENTIONS:
Drug: Vaenicline oral tablet 1 mg, then OC-01 (varenicline solution) nasal spray 0.12 mg — Cross over bioavailability study
  Other Names: varenicline
  Arms: Varenicline oral tablet 1mg, then OC-01 (varenicline solution) nasal spray 0.12 mg
Drug: OC-01 (varenicline solution) nasal spray 0.12 mg then Varenicline oral tablet 1 mg — Cross over bioavailability study
  Other Names: varenicline
  Arms: OC-01 (varenicline solution) nasal spray 0.12 mg, then Varenicline oral tablet 1 mg

SUMMARY:
To assess the relative bioavailability of varenicline administered intranasally at its highest intended clinical strength compared to varenicline administered orally at its highest oral tablet strength.

DETAILED DESCRIPTION:
This study was a Phase 1, open-label, randomized, 2-way crossover study to evaluate the relative bioavailability of OC-01 (varenicline) Nasal Spray compared to varenicline administered orally as varenicline oral tablet. Approximately 22 healthy volunteer subjects between 18-65 years of age meeting all other study eligibility criteria were randomized (Treatment Period 1) to receive an intranasal dose of 0.12 mg OC-01 (50 µL spray of 0.06 mg into each nostril) or a single 1 mg oral dose of varenicline oral tablet. Both administrations were delivered while subject is in an overnight fasted state. Subjects then returned at least 14 days later (Treatment Period 2) to receive the alternate dose of varenicline that was delivered at Treatment Period 1. Again, this delivery was performed while subject was in an overnight fasted state.

Participants who terminated early during the application period were asked to complete safety assessments (if the participants agree) prior to study exit. Participants who were terminated early from the study were not replaced.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index between 18.0 and 32.0 kg/m2, inclusive.
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, ECG and laboratory tests.
* Have provided verbal and written informed consent
* If a female of childbearing potential who is not using an acceptable means of birth control (acceptable methods of contraception include: hormonal - oral, implantable, injectable, or transdermal contraceptives, mechanical - spermicide in conjunction with a barrier such as a diaphragm or condom, IUD, or surgical sterilization of partner), have a negative urine pregnancy test at the Screening Visit.

Exclusion Criteria:

* Have had nasal or sinus surgery (including history of application of nasal cautery) or significant trauma to these areas.
* Have a vascularized polyp, severely deviated septum, chronic recurrent nosebleeds, or severe nasal airway obstruction as confirmed by intranasal examination at the Screening Visit.
* Any contraindication to varenicline according to the applicable label.
* Have severe renal impairment (estimated creatinine clearance less than 30mL per minute)
* Have current concomitant use of snuff, chewing tobacco, e-cigarettes or cigarettes/cigars during the study
* Have any condition or history that, in the opinion of the investigator, may interfere with study compliance, outcome measures, safety parameters, and/or the general medical condition of the subject
* Be a female who is pregnant, nursing an infant, or planning a pregnancy at the Screening Visit. Be a woman of childbearing potential who is not using an acceptable means of birth control; acceptable methods of contraception include: hormonal - oral, implantable, injectable, or transdermal contraceptives; mechanical - spermicide in conjunction with a barrier such as a diaphragm or condom; IUD; or surgical sterilization of partner.
* Be currently enrolled in an investigational drug or device study or have used an investigational drug or device within 30 days prior to the Screening Visit.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-08-26 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2019-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Nau, PhD, Study Director — Oyster Point Pharma, Inc.
Locations (1):
- United States, Miami Florida, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nau J, Wyatt DJ, Rollema H, Crean CS. A Phase I, Open-label, Randomized, 2-Way Crossover Study to Evaluate the Relative Bioavailability of Intranasal and Oral Varenicline. Clin Ther. 2021 Sep;43(9):1595-1607. doi: 10.1016/j.clinthera.2021.07.020. Epub 2021 Aug 27. PMID 34456060

RESULTS

PARTICIPANT FLOW:
Groups:
- Varenicline Oral Tablet 1 mg, Then OC-01 (Varenicline) Nasal 0.12 mg: Treatment sequence A: single oral dose of 1 mg varenicline tablet, washout for 14 days, then treatment sequence B intranasal dose of 0.12 mg OC-01 nasal spray.
- OC-01 (Varenicline Solution) Nasal Spray 0.12 mg, Then Varenicline Oral Tablet 1 mg: Treatment sequence B intranasal dose of 0.12 mg OC-01 nasal spray, washout for 14 days, then treatment sequence A: single oral dose of 1 mg varenicline tablet.
Period: Overall Study
Arm/Group | Varenicline Oral Tablet 1 mg, Then OC-01 (Varenicline) Nasal 0.12 mg | OC-01 (Varenicline Solution) Nasal Spray 0.12 mg, Then Varenicline Oral Tablet 1 mg
Started | 11 | 11
Completed | 11 | 10
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- OC-01 (Varenicline Solution) Nasal Spray 0.12 mg Then Varenicline Oral Tablet 1 mg: Treatment sequence A: single oral dose of 1 mg varenicline tablet, washout for 14 days, then treatment sequence B: intranasal dose of 0.12 mg OC-01 nasal spray.
- Varenicline Oral Tablet 1 mg Then OC-01 (Varenicline Solution) Nasal Spray 0.12 mg: Treatment sequence B: intranasal dose of 0.12 mg OC-01 nasal spray, washout for 14 days, then treatment sequence A: single oral dose of 1 mg varenicline tablet.
- Total: Total of all reporting groups
Arm/Group | OC-01 (Varenicline Solution) Nasal Spray 0.12 mg Then Varenicline Oral Tablet 1 mg | Varenicline Oral Tablet 1 mg Then OC-01 (Varenicline Solution) Nasal Spray 0.12 mg | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Customized [Mean (Standard Deviation); unit: years]
  age | 39.5 (10.6) | 44.5 (14.0) | 42.0 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 7 | 10
  Male | 8 | 4 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 9 | 19
  Not Hispanic or Latino | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: AUC0-t
Description: Area under the curve from predose (time 0), 0.083, 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, and 120 hours post dose.
Time Frame: Blood samples were taken predose (time 0), 0.083, 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, and 120 hours post dose.
Population: Pharmacokinetic analysis set. Subjects who completed both periods and have sufficient data to calculate AUC0-t were included.
Measure: Mean (Standard Deviation); unit: h*ng/ml
Groups:
- Varenicline Oral Tablet 1 mg: OC-01 0.12 mg was administered intranasally 50 ul into each nostril in a fasted state Vaenicline oral tablet 1 mg, then OC-01 (varenicline solution) nasal spray 0.12 mg
- OC-01 (Varenicline) Nasal Spray 0.12 mg: Varenicline oral tablet 1mg was administered orally in a fasted stated with 200 ml water OC-01 (varenicline solution) nasal spray 0.12 mg then Varenicline oral tablet 1 mg.
Arm/Group | Varenicline Oral Tablet 1 mg | OC-01 (Varenicline) Nasal Spray 0.12 mg
Number analyzed (Participants) | 16 | 16
h*ng/ml | 4.49 (3.42) | 98.74 (25.49)

2. Primary Outcome: AUC0-inf
Description: AUC0-inf taken at predose (time 0), 0.083, 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, and 120 hours post dose.
Time Frame: as for outcome 1
Population: Pharmacokinetic analysis set. Subjects who completed both periods and have sufficient data to calculate AUC0-∞
Measure: Mean (Standard Deviation); unit: h*ng/mL
Groups:
- OC-01 (Varenicline) Nasal Spray 0.12 mg: OC-01 0.12 mg was administered intranasally 50 ul into each nostril in a fasted state
  Vaenicline oral tablet 1 mg, then OC-01 (varenicline solution) nasal spray 0.12 mg
- Varenicline Oral Tablet 1 mg: Varenicline oral tablet 1mg was administered orally in a fasted stated with 200 ml water
  OC-01 (varenicline solution) nasal spray 0.12 mg then Varenicline oral tablet 1 mg
Arm/Group | OC-01 (Varenicline) Nasal Spray 0.12 mg | Varenicline Oral Tablet 1 mg
Number analyzed (Participants) | 16 | 16
h*ng/mL | 8.3 (4.09) | 102.83 (16.82)

3. Primary Outcome: Cmax
Description: Cmax taken at predose (time 0), 0.083, 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, and 120 hours post dose.
Time Frame: as for outcome 1
Population: Pharmacokinetic analysis set. Subjects who completed both periods and have sufficient data to calculate Cmax were included.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | OC-01 (Varenicline) Nasal Spray 0.12 mg | Varenicline Oral Tablet 1 mg
Number analyzed (Participants) | 16 | 16
ng/ml | 0.34 (0.13) | 4.63 (0.93)

4. Primary Outcome: Tmax
Description: Tmax taken at predose (time 0), 0.083, 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, and 120 hours post dose.
Time Frame: as for outcome 1
Measure: Median (Full Range); unit: h
Arm/Group | OC-01 (Varenicline) Nasal Spray 0.12 mg | Varenicline Oral Tablet 1 mg
Number analyzed (Participants) | 16 | 16
h | 2.0 [0.3 to 3.0] | 3 [1 to 6]

5. Other Pre Specified Outcome: Creatine Shift From Normal at Baseline to Abnormal After 2 Hours Post-treatment
Description: Creatine shift from baseline to 2 hours post treatment. Elevated creatinine may indicate impaired kidney function.
Time Frame: Baseline to 2 hours post treatment
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Varenicline Oral Tablet 1mg, Then OC-01 (Varenicline Solution) Nasal Spray 0.12 mg | OC-01 (Varenicline Solution) Nasal Spray 0.12 mg, Then Varenicline Oral Tablet 1 mg
Number analyzed (Participants) | 22 | 21
Participants | 3 | 3

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from the first dose of study drug administration until the final study visit (60 days).
Description: In the Varenicline Oral Tablet 1 mg, Then OC- 01 (Varenicline) Nasal Spray 0.12 mg arm, 1 subject withdrew after receiving the Varenicline oral tablet and before receiving the OC-01 (varenicline) nasal spray
Groups:
- OC- 01 (Varenicline) Nasal Spray 0.12 mg: OC- 01 (varenicline) nasal spray 0.12 mg
- Varenicline Oral Tablet 1 mg: Varenicline oral tablet 1 mg
Arm/Group | OC- 01 (Varenicline) Nasal Spray 0.12 mg | Varenicline Oral Tablet 1 mg
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/22
Other Adverse Events (participants affected / at risk) | 13/21 | 9/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OC- 01 (Varenicline) Nasal Spray 0.12 mg (N=21) | Varenicline Oral Tablet 1 mg (N=22)
nausea (Gastrointestinal disorders) | 0 | 5
vomiting (Gastrointestinal disorders) | 0 | 4
somnolence (Nervous system disorders) | 1 | 3
Sneezing (Respiratory, thoracic and mediastinal disorders) | 7 | 0
cough (Respiratory, thoracic and mediastinal disorders) | 6 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1
Chills (General disorders) | 0 | 1
Feeling cold (General disorders) | 0 | 1
Scratch (Injury, poisoning and procedural complications) | 0 | 1
Head discomfort (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 8
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal pruritus (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-07-13): https://cdn.clinicaltrials.gov/large-docs/46/NCT04072146/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-09): https://cdn.clinicaltrials.gov/large-docs/46/NCT04072146/SAP_001.pdf